CLINICAL TRIAL: NCT00111046
Title: Post-Operative Pain Relief Following Insertion of Radioactive Plaque for Choroidal Melanoma: Randomised Control Trial of Tramadol Vs Ibuprofen: A Pilot Study
Brief Title: Pain Relief - Tramadol Versus Ibuprofen
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Liverpool University Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2K/261; R&D 1931
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2005-11-10 (Estimated); Status verified 2005-05

CONDITIONS: Choroidal Melanoma; Melanoma; Eye Neoplasms
Keywords: Pain Relief; Choroidal melanoma; plaque radiotherapy
MeSH Terms: conditions — Uveal Melanoma; Melanoma; Eye Neoplasms | interventions — Ibuprofen; Tramadol

INTERVENTIONS:
Drug: Ibuprofen
Drug: Tramadol

SUMMARY:
The purpose of this study is to assess post operative pain following the insertion of radioactive plaque for choroidal melanoma in patients after receiving either ibuprofen or tramadol.

DETAILED DESCRIPTION:
Patients with choroidal melanomas who are offered ruthenium plaque radiotherapy have their plaque sutured to the sclera under general anaesthesia. The plaque is removed in a few days after delivering the required radioactive dosage to the tumour. While the plaque is in situ, patients require analgesia. The management of post-operative pain is generally not considered a high priority, more importance being given to the regression of the melanoma.

This is indicated by the lack of any study addressing this aspect of care. The failure of patients in general, to complain, may perhaps be due to them having accepted that some degree of pain following 'major surgery for a malignant ocular condition' is the norm.

As per current protocol, ibuprofen is being prescribed, unless contraindicated. Although many are comfortable, others request additional analgesics. Most opioid analgesics provide better pain relief but are associated with nausea, vomiting, constipation and respiratory depression.

Tramadol is an opioid analgesic that is reported to have less of the above mentioned side affects.

Comparisons: To compare the analgesic effect of oral tramadol versus ibuprofen in such patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients that are admitted for undergoing plaque radiotherapy for choroidal melanoma would be approached to participate in this study.
* They should be adults who are of a sound frame of mind to give an informed consent to participate.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients of unsound mind not capable of giving informed consent
* Active peptic ulcer disease, asthma, renal dysfunction, warfarin therapy, hypothyroidism history of epilepsy, pregnancy, breastfeeding and hypersensitivity to either products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-02; Study Completion 2004-02

PRIMARY OUTCOMES:
Compare levels of pain

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Damato, Principal Investigator — Royal Liverpool University Hospital
Locations (1):
- Royal Liverpool University Hospital, Liverpool, Merseyside, United Kingdom